CLINICAL TRIAL: NCT05507567
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2a Study To Assess the Safety, Tolerability and Prophylactic Antiviral Activity of Neumifil Against Influenza, Via a Human Viral Challenge Model in Healthy Adult Participants
Brief Title: Safety, Tolerability and Prophylactic Antiviral Activity of Neumifil Against Influenza Via a Human Viral Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pneumagen Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PNG-NMF-201
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Influenza Viral Infections
Keywords: Influenza; Human Challenge; Prophylaxis
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neumifil multiple dose prophylactic treatment (Experimental): Neumifil intranasal spray administered as 3 single daily doses prior to viral challenge
  Interventions: Drug: Neumifil
- Neumifil single dose prophylactic treatment (Experimental): Neumifil intranasal spray administered as a single dose and blinded by placebo administered as two single daily doses. All administrations completed prior to viral challenge
  Interventions: Drug: Neumifil; Drug: Placebo
- Placebo (Placebo Comparator): Intranasal spray administered as 3 single daily doses prior to viral challenge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neumifil — Liquid for intranasal spray administration
  Arms: Neumifil multiple dose prophylactic treatment; Neumifil single dose prophylactic treatment
Drug: Placebo — Liquid for intranasal spray administration
  Arms: Neumifil single dose prophylactic treatment; Placebo

SUMMARY:
Study to assess the efficacy and safety of a multiple dose regimen and a single dose regimen of intranasal Neumifil, administered prior to challenge with Influenza virus in healthy adult participants

DETAILED DESCRIPTION:
This is a single-centre, randomized, double-blind, placebo-controlled study in healthy adult participants to assess the pre-exposure prophylactic antiviral activity of Neumifil via a human viral challenge model.

Participants will enter the quarantine unit on Day -4.

Participants will be randomized to receive either active (single dose), active (multiple dose) or placebo in a 3:3:4 ratio followed by influenza viral challenge on Day 0.

Participants will leave the unit on Day 8, provided that no virus is detected by a qualitative virus antigen test and the participant has no clinically significant symptoms. A final follow-up will be performed on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the participant and the investigator obtained before any assessment is performed.
2. Adult male or female aged between 18 and 55 years old, inclusive, on the day prior to signing the consent form.
3. A total body weight ≥50 kg and body mass index (BMI) ≥18 kg/m2 and ≤35kg/m2.
4. In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that that will interfere with participant safety, as defined by medical history, physical examination, (including vital signs), ECG, and routine laboratory tests as determined by the investigator.
5. Participants will have a documented medical history either prior to entering the study or following medical history review with the study physician at screening.
6. Agree to use highly effective contraception
7. Serosuitable for the challenge virus

Exclusion Criteria:

1. History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract (URT, LRT) infection within 4 weeks prior to the first study visit.
2. Any history or evidence of any clinically significant or currently active cardiovascular, respiratory, dermatological, gastrointestinal, endocrinological, haematological, hepatic, immunological (including immunosuppression), metabolic, urological, renal, neurological, or psychiatric disease and/or other major disease that, in the opinion of the investigator, may interfere with a participant completing the study and necessary investigations. Includes a history of depression or anxiety.
3. Any participants who have smoked ≥ 10 pack years at any time.
4. Females who are pregnant or breastfeeding
5. Any history of anaphylaxis or history of severe allergic reactions to any foods, drugs, insect bites or stings or any known allergy to tetracycline antibiotics.
6. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
7. a) Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and, in particular, any of the nasal assessments or viral challenge b) Any evidence of nasal inflammation or nasal polyps within the last month c) Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalised due to epistaxis on any previous occasion.

   d) Any nasal or sinus surgery within 3 months of the first study visit. Prior or Concomitant Medications and Assessments
8. a) Evidence of vaccinations within the 4 weeks prior to the planned date of first dosing with IMP.

   b) Intention to receive any vaccination(s) before the last day of follow-up (with the exception of vaccinations recommended for COVID19 as defined by Medicines and Healthcare Regulatory Agency (MHRA)/government vaccination guidelines). No travel restrictions apply after the Day 28 (±3 days) follow-up visit.

   c) Receipt of influenza vaccine (or another IMP relating to treatment of influenza) in the last 6 months prior to the planned date of viral challenge OR a diagnosis of influenza or influenza-like illness confirmed by a physician within the last 2 months prior to screening.
9. Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 3 months prior to the planned date of first dosing with IMP or planned during the 3 months after the final follow-up visit.
10. a) Receipt of any investigational drug within 3 months (or 5 half-lives of the IMP used in the other study, whichever is greater), prior to the planned date of first dosing with IMP.

    b) Receipt of 3 or more investigational drugs within the previous 12 months prior to the planned date of first dosing with IMP.

    c) Prior inoculation with a virus from the same virus-family as the challenge virus.

    d) Prior participation in another human viral challenge study with a respiratory virus in the preceding 3 months.
11. Use or anticipated use during the conduct of the study of concomitant medications
12. Confirmed positive test for drugs of misuse and cotinine on first study visit

13 Recent history or presence of alcohol addiction, or excessive use of alcohol

14. A FEV1 <80%, a FVC <80% predicted, or an FEV1/FVC ratio <0.7. 15. Positive HIV, hepatitis B virus, or hepatitis C virus test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.com
Locations (1):
- hVIVO Services Limited, London, United Kingdom

REFERENCES:
- [Derived] Kitson G, Byford M, Cass L, Howat D, Kohn B, Bisquera A, Catchpole A, Noulin N, Thomson D. A Phase II, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of HEX17, a Novel Broad-Spectrum Antiviral Drug, in a Controlled Human Infection Model of Influenza Challenge. Infect Dis Ther. 2025 Aug;14(8):1697-1714. doi: 10.1007/s40121-025-01179-2. Epub 2025 Jul 2. PMID 40593264

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following screening (Day -93 to Day -5), this study was conducted with an inpatient phase (Day -4 to Day 8) and an outpatient follow-up on Day 28 (plus or minus 3 days). During the inpatient quarantine phase, participants received Neumifil or placebo according to the randomisation on Day -3, Day -2 and Day -1, and then received Influenza Challenge Virus on Day 0. The study was conducted at one site in the UK between 12 August 2022 and 03 May 2023.
Groups:
- Neumifil Single Dose Prophylactic Treatment: Neumifil intranasal spray administered as a single dose on Day -3 and blinded by placebo administered as two single daily doses. All administrations completed prior to viral challenge
  Neumifil: Liquid for intranasal spray administration
  Placebo: Liquid for intranasal spray administration
Period: Randomised and Received Challenge Virus
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo
Started | 32 | 31 | 41
Completed | 30 | 31 | 40
Not Completed | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Did not complete quarantine | 1 | 0 | 0
Period: From Challenge Virus to End of Study
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo
Started | 30 | 31 | 40
Completed | 30 | 29 | 40
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Total
Number analyzed (Participants) | 32 | 31 | 41 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.22 (6.79) | 30.32 (7.06) | 31.05 (8.82) | 30.88 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 14 | 32
  Male | 23 | 22 | 27 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 31 | 29 | 39 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 5 | 4 | 9
  White | 21 | 22 | 33 | 76
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 6 | 3 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 31 | 41 | 104

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Symptomatic Influenza Infection
Description: Number of subjects with quantifiable viral shedding on 2 consecutive days AND with any symptom score of grade 2 or greater at a single time point.
  Viral shedding was measured by RT-qPCR. Eleven symptoms were assessed by questionnaire and were graded on a scale of 0-3 (grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; grade 3: quite bothersome most or all of the time, and it stops me participating in activities).
Time Frame: Day 1 to Day 8
Population: Per Protocol population (participants who received all doses, challenge virus and completed quarantine up to Day 8)
Measure: Count of Participants; unit: Participants
Groups:
- Neumifil Single Dose Prophylactic Treatment: Neumifil intranasal spray administered as a single daily dose on Day -3 prior to viral challenge
- Placebo: Placebo intranasal spray administered as 3 single daily doses prior to viral challenge
- Pooled Neumifil Groups: Pooled groups:Neumifil intranasal spray administered prior to viral challenge
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 30 | 29 | 40 | 59
Participants | 6 | 6 | 16 | 12
Statistical Analysis 1: Comparison: Placebo vs Pooled Neumifil Groups; A priori primary analysis group; Test type: Other; p = 0.0331, Chi-squared

2. Primary Outcome: Severity of Symptoms
Description: Change in Peak Total Symptom Score (TSS) as measured by graded symptom scoring system collected 3 times daily; symptom questionnaire was graded on a scale of 0-3 (grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; grade 3: quite bothersome most or all of the time, and it stops me participating in activities).Lower score means better outcome. The range was 0 to 33.
Time Frame: Day 1 to Day 8
Population: Per Protocol population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 30 | 29 | 40 | 59
Scores on a scale | 3.00 [0.0 to 16.0] | 1.00 [0.0 to 12.0] | 3.00 [0.0 to 17.0] | 2.00 [0.0 to 16.0]
Statistical Analysis 1: Comparison: Placebo vs Pooled Neumifil Groups; Test type: Other; p = 0.1427, Wilcoxon (Mann-Whitney) — Hodges-Lehmann (H-L) estimation; 1-sided Wilcoxon rank-sum

3. Secondary Outcome: Area Under the Curve (AUC) Over Time of Total Symptom Score (TSS)
Description: Participants completed a self-assessment symptom score 3 times daily, graded on a scale of 0-3 (grade 0: no symptoms; grade 1: just noticeable; grade 2: clearly bothersome from time to time but does not interfere with me doing my normal daily activities; grade 3: quite bothersome most or all of the time, and it stops me participating in activities).Lower score means better outcome. Range 0 to 33
Time Frame: Day 1 to Day 8
Population: Per Protocol population
Measure: Median (Full Range); unit: (Units on a scale)*day
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 30 | 29 | 40 | 59
(Units on a scale)*day | 4.05 [0.0 to 47.7] | 0.11 [0.0 to 25.8] | 3.73 [0.0 to 50.0] | 2.44 [0.0 to 47.7]
Statistical Analysis 1: Comparison: Placebo vs Pooled Neumifil Groups; Test type: Other; p = 0.1307, Wilcoxon (Mann-Whitney) — H-L estimation; 1-sided Wilcoxon rank-sum

4. Secondary Outcome: Viral Shedding Over Time
Description: Measurement of influenza viral load (VL) area under the curve (VL-AUC) of quantifiable measurements by RT-qPCR in nasal samples.
  The AUC is expressed as the log to the base 10 copies in a mL of nasal fluid multiplied by the time in days [(log10 copies/mL)*day]. The higher the viral load AUC, by PCR, the worse the outcome.
Time Frame: Day 1 (pm) to Day 8 (am)
Population: Per Protocol Population
Measure: Median (Full Range); unit: (log10 copies/mL)*day
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 30 | 29 | 40 | 59
(log10 copies/mL)*day | 9.96 [6.3 to 40.2] | 8.60 [6.3 to 39.0] | 17.24 [6.3 to 44.8] | 9.39 [6.3 to 40.2]
Statistical Analysis 1: Comparison: Placebo vs Pooled Neumifil Groups; Test type: Other; p = 0.0382, Wilcoxon (Mann-Whitney) — H-L estimation; 1-sided Wilcoxon rank-sum

5. Secondary Outcome: Viral Shedding Over Time
Description: Measurement of influenza viral load (VL) in nasal samples over time (VL-AUC) measured by viral culture. Nasal secretions were cultured and the Tissue Culture Infectious Dose (TCID50) calculated. The AUC of log to the base 10 of the TCID50 in each mL of nasal secretions, multiplied by the time in days [(log10 TCID50/mL)*day] was calculated. The higher the viral load AUC by culture, the worse the outcome.
Time Frame: Day 1 (pm) to Day 8 (am)
Population: Per Protocol population (one participant in the placebo group had a missing value)
Measure: Median (Full Range); unit: (log10 TCID50/mL)*day
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 30 | 29 | 39 | 59
(log10 TCID50/mL)*day | 3.29 [3.2 to 15.7] | 3.30 [3.2 to 18.0] | 4.79 [3.2 to 17.9] | 3.30 [3.2 to 18.0]
Statistical Analysis 1: Comparison: Placebo vs Pooled Neumifil Groups; Test type: Other; p = 0.0110, Wilcoxon (Mann-Whitney) — H-L estimation; 1-sided Wilcoxon rank-sum

6. Secondary Outcome: Weight of Nasal Discharge
Description: Measurement of total weight of mucus produced by participants. The total weight of used tissues was measured to assess the weight of mucus produced. The greater the weight of the tissues the more mucus produced and the worse the outcome.
Time Frame: Day 1 (am) to Day 8 (am)
Population: Per Protocol population (Data not available for all participants)
Measure: Median (Full Range); unit: grams
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 23 | 24 | 35 | 47
grams | 5.24 [0.0 to 83.2] | 0.26 [0.0 to 54.2] | 2.74 [0.0 to 43.7] | 0.97 [0.0 to 83.2]

7. Secondary Outcome: Nasal Discharge
Description: The number of tissues used by participants were counted. The greater the number of tissues used the worse the outcome.
Time Frame: Day 1 (am) to Day 8 (am)
Population: Per Protocol population (Data not available for all participants)
Measure: Median (Full Range); unit: sum of number of tissues
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo | Pooled Neumifil Groups
Number analyzed (Participants) | 25 | 25 | 35 | 50
sum of number of tissues | 14.00 [0.0 to 144.0] | 2.00 [0.0 to 88.0] | 7.00 [0.0 to 52.0] | 5.5 [0.0 to 144.0]

8. Secondary Outcome: Adverse Events, Solicited
Description: Number of participants reporting a solicited adverse event during the treatment period of IMP
Time Frame: From intake of first dose of IMP (Day -3) up to 12 hours post the last IMP dose (Day -1)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo
Number analyzed (Participants) | 32 | 31 | 41
Participants | 29 | 22 | 29

9. Secondary Outcome: Adverse Events, Unsolicited
Description: Number of participants reporting treatment emergent adverse events, unsolicited
Time Frame: From intake of first dose of IMP on Day -3 to Day 28
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo
Number analyzed (Participants) | 32 | 31 | 41
Participants | 9 | 8 | 17

ADVERSE EVENTS:
Time Frame: From the intake of the first dose of IMP on Day -3 to Day 28
Description: Unsolicited Treatment Emergent Adverse Events were collected by open and non-leading verbal questioning from Day -3 to Day 28.
  Solicited adverse events were collected using participant completed questionnaires 1 hour and 12 hours after each dose of study medication from Day -3 to Day -1.
Groups:
- Neumifil Single Dose Prophylactic Treatment: Neumifil intranasal spray administered as a single daily dose on Day -3 and blinded by placebo administered as two single daily doses. All administrations completed prior to viral challenge
  Neumifil: Liquid for intranasal spray administration
  Placebo: Liquid for intranasal spray administration
Arm/Group | Neumifil Multiple Dose Prophylactic Treatment | Neumifil Single Dose Prophylactic Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/41
Other Adverse Events (participants affected / at risk) | 30/32 | 25/31 | 34/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neumifil Multiple Dose Prophylactic Treatment (N=32) | Neumifil Single Dose Prophylactic Treatment (N=31) | Placebo (N=41)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) — Indicates events were unsolicited
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Indicates events were unsolicited
Tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Indicates events were unsolicited
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave biphasic (Investigations) | 0 (0) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Indicates events were unsolicited
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Indicates events were unsolicited
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Indicates events were unsolicited
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — Indicates events were unsolicited
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Indicates events were unsolicited
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Indicates events were unsolicited
Bleeding from the nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (6) — Indicates events were solicited
Burning sensation or sensation of heat/hotness in the nose (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (7) | 5 (8) — Indicates events were solicited
General irritation in the nose (Respiratory, thoracic and mediastinal disorders) | 16 (40) | 12 (26) | 16 (32) — Indicates events were solicited
Marked change in sense of smell or taste (Nervous system disorders) | 3 (6) | 1 (1) | 1 (2) — Indicates events were solicited
Pain or stinging in the nose (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 8 (11) | 6 (10) — Indicates events were solicited
Sensation of needing to blow your nose (Respiratory, thoracic and mediastinal disorders) | 22 (70) | 14 (30) | 12 (28) — Indicates events were solicited
Sneezing (Respiratory, thoracic and mediastinal disorders) | 18 (40) | 11 (18) | 15 (30) — Indicates events were solicited
Unpleasant taste (Gastrointestinal disorders) | 12 (27) | 8 (10) | 13 (22) — Indicates events were solicited

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT05507567/Prot_SAP_000.pdf